CLINICAL TRIAL: NCT03342690
Title: DRUG USE INVESTIGATION OF SELARA(REGISTERED). TABLETS(AN INVESTIGATION FOR CHRONIC HEART FAILURE)
Brief Title: Drug Use Investigation of Selara Tablets (an Investigation for Chronic Heart Failure)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6141122
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Results first posted 2021-06-28 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Chronic Heart Failure
Keywords: Selara; Chronic Heart Failure
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eplerenone: Patients with CHF receiving Selara (eplerenone)
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — In adults, usually, administer the initial dose of 25 mg once daily according to the patient's serum potassium level and conditions, increase dosage up to 50 mg once daily after 4 week; patients with moderate renal impairment should start with 25 mg every other day and the maximum dosage should be 25 mg once daily.
  Also, dose should be reduced or interrupted according to serum potassium level and patient's conditions.
  Other Names: Selara

SUMMARY:
Secondary Data Collection Study; Safety And Effectiveness Of Selara Under Japanese Medical Practice

DETAILED DESCRIPTION:
This study will be conducted under the central registration system until the number of subjects who meet the conditions for registration reaches the target number of subjects. The patients will be observed up until Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom treatment with this drug is for CHF. The indications at approval for this drug are as follows. When using this drug, refer to the latest package insert of this drug.

Exclusion Criteria:

* Patients who were previously registered for this study. Patients who received eplerenone within the past three months regardless of the reason for use.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who meet the inclusion criteria and who were registered to this study within 14 days including the start date of treatment with this product will be subjects for this study
Sampling Method: Probability Sample
Enrollment: 1165 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country Office, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6141122

RESULTS

PARTICIPANT FLOW:
Groups:
- Selara Tablets (Eplerenone): Participants who received Selara as indicated in the approved local product document were observed for a period of 52 weeks. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Selara Tablets (Eplerenone)
Started | 1164
Completed | 1139
Not Completed | 25
Not completed — Missing Information | 9
Not completed — Protocol Violation | 16

BASELINE CHARACTERISTICS:
Population: A total of 1165 participants were enrolled in this study. Of the 1164 participants who completed the study, 25 participants were excluded from the safety analysis set due to the following reasons: protocol violation (16 participants), and no adverse event information (no visit after first day of treatment or unknown) (9 participants).
Arm/Group | Selara Tablets (Eplerenone)
Number analyzed (Participants) | 1139
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 219
  ≥65 years | 920
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 516
  Male | 623
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Estimated creatinine clearance (eCLCr) [Number; unit: Participants] — The Cockcroft & Gault formula was used to eCLCr.
  Participants
    <30 mL/min | 92
    ≥30 mL/min and <50 mL/min | 316
    ≥50 mL/min | 524
    Unknown | 207

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reactions in Chronic Heart Failure Participants With Moderate Renal Impairment
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Selara in a chronic heart failure participant with moderate renal impairment (≥30 mL/min and <50 mL/min in eCLCr) who received Selara. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Selara was assessed by the physician.
Time Frame: 52 weeks from the start date
Population: The safety analysis set comprised of chronic heart failure participants who satisfied the inclusion criteria and had received Selara at least once. Of the participants included in the safety analysis set (n=1139), 316 participants had moderate renal impairment (≥30 mL/min and <50 mL/min in eCLCr).
Measure: Number; unit: Percentage of Participants
Arm/Group | Selara Tablets (Eplerenone)
Number analyzed (Participants) | 316
Percentage of Participants
  ADR | 9.49
  Serious ADR | 1.58

2. Secondary Outcome: Percentage of Participants With Adverse Drug Reactions in Chronic Heart Failure Participants
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Selara in a chronic heart failure participant who received Selara. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Selara was assessed by the physician.
Time Frame: 52 weeks from the start date
Population: The safety analysis set comprised of chronic heart failure participants who satisfied the inclusion criteria and had received Selara at least once.
Measure: Number; unit: Percentage of Participants
Arm/Group | Selara Tablets (Eplerenone)
Number analyzed (Participants) | 1139
Percentage of Participants
  ADR | 5.97
  Serious ADR | 0.79

3. Secondary Outcome: The Number of Deaths (Overall Deaths)
Description: Overall deaths were described with the number of deaths from any cause at the time of 52 weeks after the start of administration, regardless of the treatment status (completed or discontinued).
Time Frame: 52 weeks from the start date
Population: The efficacy analysis set comprised of chronic heart failure participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once.
Measure: Number; unit: Participants
Arm/Group | Selara Tablets (Eplerenone)
Number analyzed (Participants) | 1139
Participants | 44

4. Secondary Outcome: The Number of Deaths (Cardiovascular Deaths)
Description: Cardiovascular deaths were described with the number of deaths defined as any death due to cardiac failure, myocardial infarction, arrhythmia (atrial fibrillation, atrial flutter, arrhythmia supraventricular, or ventricular arrhythmia), stroke or cerebrovascular attack, and other causes related to cardiovascular system at the time of 52 weeks after the start of administration, regardless of the treatment status (completed or discontinued).
Time Frame: 52 weeks from the start date
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Selara Tablets (Eplerenone)
Number analyzed (Participants) | 1139
Participants | 15

5. Secondary Outcome: The Overall Mortality Rate
Description: The overall mortality rate was calculated by the incidence of all-cause death per observation time based on the person-year method (the number of deaths in 100 person-year).
Time Frame: 52 weeks from the start date
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: events per 100 patient-year
Arm/Group | Selara Tablets (Eplerenone)
Number analyzed (Participants) | 1139
events per 100 patient-year | 4.4 [3.2 to 6.0]

6. Secondary Outcome: The Cardiovascular-related Mortality Rate
Description: The cardiovascular-related mortality rate was calculated by the incidence of cardiovascular-related death per observation time based on the person-year method (the number of deaths in 100 person-year).
  Cardiovascular deaths were defined as any death due to cardiac failure, myocardial infarction, arrhythmia (atrial fibrillation, atrial flutter, arrhythmia supraventricular, or ventricular arrhythmia), stroke or cerebrovascular attack, and other causes related to cardiovascular system at the time of 52 weeks after the start of administration, regardless of the treatment status (completed or discontinued).
Time Frame: 52 weeks from the start date
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: events per 100 patient-year
Arm/Group | Selara Tablets (Eplerenone)
Number analyzed (Participants) | 1139
events per 100 patient-year | 1.5 [0.8 to 2.5]

ADVERSE EVENTS:
Time Frame: 52 weeks from the start date
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | Selara Tablets (Eplerenone)
All-Cause Mortality (participants affected / at risk) | 44/1139
Serious Adverse Events (participants affected / at risk) | 103/1139
Other Adverse Events (participants affected / at risk) | 121/1139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selara Tablets (Eplerenone) (N=1139)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 5
Right ventricular failure (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 7
Angina pectoris (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 3
Ventricular tachycardia (Cardiac disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 15
Atrial flutter (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 6
Deafness neurosensory (Ear and labyrinth disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Hypothermia (General disorders) | 2
Amyloidosis (Immune system disorders) | 1
Influenza (Infections and infestations) | 1
Infective spondylitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Pneumonia pneumococcal (Infections and infestations) | 1
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
Embolic stroke (Nervous system disorders) | 2
Brain stem infarction (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 4
Renal impairment (Renal and urinary disorders) | 2
Postrenal failure (Renal and urinary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selara Tablets (Eplerenone) (N=1139)
Anaemia (Blood and lymphatic system disorders) | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Oedema (General disorders) | 3
Pyrexia (General disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Bronchitis (Infections and infestations) | 2
Parotitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Heat illness (Injury, poisoning and procedural complications) | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood potassium increased (Investigations) | 4
Blood pressure decreased (Investigations) | 9
Blood pressure increased (Investigations) | 1
Blood urea increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 16
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Carotid artery aneurysm (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Prerenal failure (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 24
Urge incontinence (Renal and urinary disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 2
Nipple pain (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03342690/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT03342690/SAP_001.pdf